CLINICAL TRIAL: NCT01219959
Title: Multi-center, Prospective, Randomized Trial to Demonstrate Improved Metabolic Control of Dianeal, Extraneal, Nutrineal (D-E-N) Versus Dianeal Only in the Treatment of Diabetic CAPD Patients
Brief Title: Dianeal, Extraneal, Nutrineal (D-E-N) Versus Dianeal Only in Diabetic Continuous Ambulatory Peritoneal Dialysis (CAPD) Patients
Acronym: EDEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51067
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease (ESRD); Diabetes; CAPD
Keywords: ESRD; Diabetes; CAPD
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus | interventions — Icodextrin; Nutrineal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-glucose Sparing (Active Comparator): Dianeal only
  Interventions: Drug: Dianeal
- Glucose Sparing (Experimental): Dianeal, Extraneal, Nutrineal
  Interventions: Drug: Dianeal, Extraneal, Nutrineal

INTERVENTIONS:
Drug: Dianeal — Dianeal 1.5% dextrose, 2.5% dextrose, 4.25% dextrose
  Arms: Non-glucose Sparing
Drug: Dianeal, Extraneal, Nutrineal — Dianeal 1.5% dextrose, 2.5% dextrose, 4.25% dextrose, Nutrineal 1.1% Amino Acids, Extraneal 7.5% Icodextrin
  Arms: Glucose Sparing

SUMMARY:
Primary Objective: To demonstrate that use of glucose sparing prescriptions, Dianeal, Extraneal, Nutrineal (D-E-N) versus Dianeal only, in diabetic (Type 1 and Type 2) Continuous Ambulatory Peritoneal Dialysis (CAPD) patients leads to improved metabolic control as measured by the magnitude of change from the baseline value in the HbA1c levels.

Secondary Objectives: To demonstrate that use of glucose-sparing Peritoneal Dialysis solutions (D-E-N versus Dianeal only) in diabetic (Type 1 and Type 2) CAPD patients leads to lower glycemic-control medication requirements, decreased incidence of severe hypoglycemic events requiring medical intervention, improved metabolic control, nutritional status, and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients 18 years of age or older
2. Diagnosis of ESRD [Glomerular Filtration Rate (GFR) ≤ 15 mL/min]
3. CAPD using only Dianeal, at least 1 exchange of 2.5% or 4.25% dextrose/day, no prescribed dry time
4. Diabetes Mellitus (Type 1 and 2)
5. HbA1c > 6.0% but ≤ 12.0%
6. Blood hemoglobin ≥ 8.0 g/dL, but ≤ 13.0 g/dL
7. Total Kt/V ≥ 1.7

Exclusion Criteria:

1. Blood Urea Nitrogen (BUN) > 95 mg/dL
2. Exposure to Extraneal within 60 days of Screening
3. Mean Arterial Pressure (MAP) ≥ 125 mm Hg, or volume depleted (MAP < 77mm Hg) at Screening
4. Peritonitis, exit-site or tunnel infection treated with antibiotics within last 30 days
5. Cardiovascular event within the last 30 days
6. Ongoing clinically significant congestive heart failure [New York Heart Association (NYHA) class III or IV]
7. Allergy to starch-based polymers, glycogen storage disease or isomaltose/maltose intolerance
8. Receiving rosiglitazone maleate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Colombia (16):
  - Nefrosalud Ltda, Armenia
  - RTS Ltda Barranquila, Barranquilla
  - RTS Ltda Soledad, Bogotá
  - Rts Ltda Ag H.U.S, Bucaramanga
  - RTS Ltda H.U.V, Cali
  - RTS Ltda STR del Valle, Cali
  - RTS Ltda Versalles, Cali
  - Renal Therapy Services (RTS) Ltda Cartagena, Cartagena
  - RTS Ltda Cucuta, Cúcuta
  - RTS Ltda Girardot, Girardot
  - Unidad Renal de Tolima, Ibagué
  - RTS Ltda Sucursal Medellin, Medellín
  - RTS Ltda Valle de Aburra, Medellín
  - RTS Ltda Sogamoso, Sogamoso
  - RTS Sucrusal Tulua, Tuluá
  - RTS Ltda Villavicencio, Villavicencio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data represented in this module is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067). Given that the glucose content of the PD solutions is similar, the pooling of the results were considered a valid method to answer the underlying research questions.
Groups:
- Non-Glucose Sparing Prescriptions: Dianeal only and/or Bieffe peritoneal dialysis (PD) solutions only
- Glucose Sparing Prescriptions: Physioneal, Extraneal, Nutrineal (PEN) used for 31998 and 34202 studies, and Dianeal, Extraneal, Nutrineal (DEN) used for 51067 study.
Period: Overall Study
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Started | 127 | 124
Completed | 120 | 101
Not Completed | 7 | 23
Not completed — Adverse Event | 6 | 14
Not completed — Physician Decision | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Renal Transplantation | 0 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The data represented in this module is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067). Given that the glucose content of the PD solutions is similar, the pooling of the results were considered a valid method to answer the underlying research questions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions | Total
Number analyzed (Participants) | 127 | 124 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.8) | 57.3 (12) | 57.65 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 64 | 123
  Male | 68 | 60 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Baseline: Asian | 41 | 42 | 83
  Baseline: Black | 1 | 0 | 1
  Baseline: Caucasian | 41 | 41 | 82
  Baseline: Hispanic | 32 | 31 | 63
  Baseline: Other | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From the Baseline Value in HbA1c at Month 3 and 6
Description: HbA1c is a specific glycohemoglobin, and adduct of glucose attached to the beta-chain terminal valine residue. Measured using a Tina-quant immunological assay suitable for samples from end stage renal disease (ESRD) patients and with icodextrin metabolites or equivalent. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: Primary Efficacy Intent-to-Treat (ITT) population included all subjects randomized with a minimum of a baseline HbA1c value determined and one PD exchange using study solution performed. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489, NCT00567398, NCT01219959.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 125 | 119
Percent Change
  Month 3 | 0.2 (1.1) | -0.6 (1.3)
  Month 6 | 0 (1.2) | -0.6 (1.5)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Month 3; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.2 to 0.9]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Month 6; Test type: Superiority; p = 0.006, ANOVA; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.1 to 0.8]

2. Secondary Outcome: Change From Baseline in Glycemic Control Medication Usage at Month 3 and 6
Description: This data used diabetic prescription drug information from insulin and oral glycemic control concomitant medications reported. Glycemic control medications classes allowed were limited to insulin, sulfonylureas, and thiazolidinediones. Subjects were provided with a paper diary on which they recorded doses of all glycemic control medications taken for 1 day prior to the Screening visit and for 8 days prior to the study visits at Month 3 and Month 6. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: Analysis used data from prescription information of concomitant medications reported. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 126 | 124
Percent Change
  Insulin: Month 3 | 3.5 (21.2) | -3.3 (16.4)
  Insulin: Month 6 | 2.9 (25.4) | -3.8 (23.9)
  Oral hypoglycemic: Month 3 | 1.3 (12.6) | 5 (51.3)
  Oral hypoglycemic: Month 6 | -0.5 (12.7) | 6.4 (52.3)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Insulin-Month 3; Test type: Superiority; p = 0.312, ANOVA; Mean Difference (Final Values) = 5, 95% CI 2-sided [-4.7 to 14.7]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Insulin-Month 6; Test type: Superiority; p = 0.342, ANOVA; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-5.0 to 14.4]

3. Secondary Outcome: Number of Severe Hypoglycemic Event Requiring Medical Intervention
Description: Severe hypoglycemia is defined by DCCT (Diabetes Control and Complications Trial) as any episode requiring external assistance to aid recovery or resulted in seizures or coma and included, as part of the definition, that the subject's blood glucose concentration had to have been documented as < 50mg/dL (<2.8mmol/L) for hypoglycemia, and/or the clinical manifestations had to have been reversed with oral carbohydrate, intramuscular glucagon, or intravenous glucose. Descriptive statistics were done, no inferential statistical analyses were performed.
Time Frame: Baseline through Month 6 (End of Study)
Population: Intent-to-Treat (ITT) population included all subjects randomized with a minimum of a baseline HbA1c value determined and one PD exchange using study solution performed. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Number; unit: events
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
events | 1 | 3

4. Secondary Outcome: Change From Baseline of Metabolic Control Determined by Lipid Profile and Triglycerides at Month 3 and 6
Description: Values for Total Cholesterol (TC), Low Density Lipoprotein Cholesterol (LDLC), High Density Lipoprotein Cholesterol (HDLC), Very Low Density Lipoprotein (VLDL), and Triglycerides are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: ITT population used. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
mmol/L
  Cholesterol: Month 3 | 0.1 (1.1) | -0.5 (1.2)
  Cholesterol: Month 6 | 0 (1.2) | -0.4 (1.2)
  LDLC: Month 3 | 0.1 (1.0) | -0.2 (1.1)
  LDLC: Month 6 | 0.1 (1.1) | -0.1 (1.2)
  HDLC: Month 3 | 0 (0.2) | 0 (0.3)
  HDLC: Month 6 | 0 (0.3) | 0 (0.3)
  VLDL: Month 3: number analyzed (Participants) | 126 | 124
  VLDL: Month 3 | -0.1 (0.9) | -0.3 (0.8)
  VLDL: Month 6: number analyzed (Participants) | 126 | 124
  VLDL: Month 6 | -0.1 (0.8) | -0.3 (0.9)
  Triglycerides: Month 3 | -0.1 (1.9) | -0.7 (1.8)
  Triglycerides: Month 6 | -0.3 (1.9) | -0.6 (1.9)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Cholesterol-Month 3; Test type: Superiority; p = 0.010, ANOVA; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.1 to 0.9]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Cholesterol-Month 6; Test type: Superiority; p = 0.073, ANOVA; Median Difference (Final Values) = 0.3, 95% CI 2-sided [0 to 0.7]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LDLC-Month 3; Test type: Superiority; p = 0.181, ANOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LDLC-Month 6; Test type: Superiority; p = 0.593, ANOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 5: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for HDLC-Month 3; Test type: Superiority; p = 0.198, ANOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0]
Statistical Analysis 6: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for HDLC-Month 6; Test type: Superiority; p = 0.298, ANOVA; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.1 to 0]
Statistical Analysis 7: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for VLDL-Month 3; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.2 to 0.6]
Statistical Analysis 8: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for VLDL-Month 6; Test type: Superiority; p = 0.003, ANOVA; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5]
Statistical Analysis 9: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Triglycerides-Month 3; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.4 to 1.3]
Statistical Analysis 10: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Triglycerides-Month 6; Test type: Superiority; p = 0.002, ANOVA; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.3 to 1.1]

5. Secondary Outcome: Change From Baseline of Metabolic Control Determined by Lipoproteins at Month 3 and 6
Description: Values for Lipoprotein A (Lp(a)), Apolipoprotein A1 (Apo A1), and Apolipoprotein B (Apo B) are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: Subset of ITT population that had evaluable data. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 119 | 120
mg/dL
  Lp(a): Month 3 (n=118,120): number analyzed (Participants) | 118 | 120
  Lp(a): Month 3 (n=118,120) | 2.3 (8.9) | 3.3 (9.8)
  Lp(a): Month 6: number analyzed (Participants) | 118 | 120
  Lp(a): Month 6 | 6.7 (15.4) | 6.8 (18)
  Apo A1: Month 3 | -2.1 (16.4) | -9.3 (17.5)
  Apo A1: Month 6 | -3.8 (17.7) | -10.5 (18.4)
  Apo B: Month 3 | 5.3 (24.2) | -8.5 (18.4)
  Apo B: Month 6 | 5.2 (25.4) | -3.6 (23.9)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Lp(a)-Month 3; Test type: Superiority; p = 0.485, ANOVA; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-8.6 to 4.1]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Lp(a)-Month 6; Test type: Superiority; p = 0.556, ANOVA; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-8.2 to 4.4]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Apo A1-Month 3; Test type: Superiority; p = 0.101, ANOVA; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-1.1 to 12.2]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Apo A1-Month 6; Test type: Superiority; p = 0.134, ANOVA; Mean Difference (Final Values) = 5, 95% CI 2-sided [-1.5 to 11.5]
Statistical Analysis 5: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Apo B-Month 3; Test type: Superiority; p = 0.004, ANOVA; Mean Difference (Final Values) = 11.4, 95% CI 2-sided [3.6 to 19.2]
Statistical Analysis 6: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Apo B-Month 6; Test type: Superiority; p = 0.030, ANOVA; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [0.8 to 15.9]

6. Secondary Outcome: Change From Baseline of Metabolic Control Determined by Insulin Action of Insulin and C-peptide at Month 3 and 6
Description: Values for Insulin and C-peptide are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: Evaluable subset of ITT population that had blood draw at baseline for these lab parameters were used. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 119 | 120
pg/mL
  Insulin: Month 3 | 70.3 (514.2) | 69.4 (809.4)
  Insulin: Month 6 | 146.3 (616) | 96.6 (1301.9)
  C-peptide: Month 3 | 340.8 (2393.7) | 70.5 (2687.2)
  C-peptide: Month 6 | 388.3 (2660.5) | 504.1 (2462.5)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Insulin-Month 3; Test type: Superiority; p = 0.655, ANOVA; Mean Difference (Final Values) = -56.5, 95% CI 2-sided [-304.6 to 191.7]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Insulin-Month 6; Test type: Superiority; p = 0.811, ANOVA; Mean Difference (Final Values) = -29.2, 95% CI 2-sided [-268.9 to 210.5]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for C-Peptide-Month 3; Test type: Superiority; p = 0.419, ANOVA; Mean Difference (Final Values) = 441.3, 95% CI 2-sided [-630.4 to 1513.1]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for C-Peptide-Month 6; Test type: Superiority; p = 0.820, ANOVA; Mean Difference (Final Values) = 121.8, 95% CI 2-sided [-927.9 to 1171.5]

7. Secondary Outcome: Change From Baseline of Metabolic Control Determined by Insulin Action of Pro-Insulin at Month 3 and 6
Description: Values for Pro-Insulin are provided. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 119 | 120
pmol/L
  Pro-Insulin: Month 3 | -1.8 (19.6) | 13 (71.3)
  Pro-Insulin: Month 6 | 3 (41.9) | 0.4 (33.5)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Pro-Insulin-Month 3; Test type: Superiority; p = 0.721, ANOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-27.5 to 19]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Pro-Insulin-Month 6; Test type: Superiority; p = 0.247, ANOVA; Mean Difference (Final Values) = 13.5, 95% CI 2-sided [-9.4 to 36.4]

8. Secondary Outcome: Number of Participants by Change From Baseline Score in Subjective Global Assessment (SGA) Class at Month 6
Description: Nutritional Status by SGA include the following: (a) Weight change over 6 months, (b) dietary history of food intake over the previous 24-hour period with a determination by the subject as to whether this was a typical or atypical diet for the subject, (c) significant and sustained gastrointestinal distress, (d) functional status, (e) metabolic stress including frequent infections, fever, peritonitis, uncontrolled diabetes and active inflammatory bowel disease. The SGA used a 7-point scale, where a decrease score in the change from baseline shows signs of increased malnourishment, and an increased score (e.g., +2) is improved nourishment. Scale: 6 - 7 = very mild risk to well-nourished; 3 - 5 = no clear sign of normal status or severe malnutrition; 1 - 2 = severely malnourished.
Time Frame: Baseline and Month 6 (End of Study)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 120 | 104
participants
  +2 Score | 1 | 2
  +1 Score | 19 | 24
  0 Score | 76 | 57
  -1 Score | 20 | 17
  -2 Score | 3 | 4
  -3 Score | 1 | 0
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimates of Ratio-Month 6; Test type: Superiority; p = 0.624, ANOVA; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.55 to 1.43]

9. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Albumin and Total Protein (Labs) at Month 3 and 6
Description: Values for Albumin and Total Protein are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
g/L
  Albumin: Month 3 | -0.1 (3.1) | -0.6 (3.6)
  Albumin: Month 6 | 0.5 (3) | -0.8 (3.9)
  Total Protein: Month 3 | 0.1 (4.3) | 0.2 (5.1)
  Total Protein: Month 6 | 0.7 (4.9) | -0.9 (6.1)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Albumin-Month 3; Test type: Superiority; p = 0.338, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.8]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Albumin-Month 6; Test type: Superiority; p = 0.029, ANOVA; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.1 to 2.5]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Total Protein-Month 3; Test type: Superiority; p = 0.817, ANOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.9 to 1.5]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Total Protein-Month 6; Test type: Superiority; p = 0.091, ANOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.2 to 2.9]

10. Secondary Outcome: Change From Baseline of Nutritional Status Determined by PNA and nPNA (Labs) at Month 3 and 6
Description: Values for Protein Nitrogen Appearance (PNA) and normalized protein nitrogen appearance (nPRNA) are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 79 | 79
g/kg/day
  PNA: Month 3 | -0.8 (14.1) | 12.8 (14.4)
  PNA: Month 6 | 1 (18.6) | 12.9 (17.5)
  nPNA: Month 3 | 0 (0.2) | 0.2 (0.2)
  nPNA: Month 6 | 0 (0.3) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for PNA-Month 3; Test type: Superiority; p = 0.127, ANOVA; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-23.3 to 2.9]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for PNA-Month 6; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-16.4 to -4.3]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for nPNA-Month 3; Test type: Superiority; p = 0.012, ANOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for nPNA-Month 6; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to -0.1]

11. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Pre-albumin (Labs) at Month 3 and 6
Description: Values for Pre-albumin are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 83 | 85
mg/dL
  Month 3 | 0.4 (7.2) | -1.9 (5.5)
  Month 6 | -1.0 (8.3) | -2.9 (5.9)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Pre-Albumin-Month 3; Test type: Superiority; p = 0.019, ANOVA; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [0.5 to 5.8]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Pre-Albumin-Month 6; Test type: Superiority; p = 0.019, ANOVA; Mean Difference (Final Values) = 3, 95% CI 2-sided [0.5 to 5.6]

12. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Drained Body Weight at Month 3 and 6
Description: Values for Drained Body Weight are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
kg
  Month 3 | -0.2 (4.5) | -0.2 (3.5)
  Month 6 | 0.2 (5.2) | -0.7 (3.3)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Drained Fat-Month 3; Test type: Superiority; p = 0.884, ANOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.9 to 3.4]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Drained Fat-Month 6; Test type: Superiority; p = 0.716, ANOVA; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3 to 4.3]

13. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Body Mass Index (BMI) at Month 3 and 6
Description: Values for BMI are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
kg/m2
  Month 3 | -0.1 (1.5) | -0.1 (1.3)
  Month 6 | 0.1 (1.9) | -0.3 (1.2)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for BMI-Month 3; Test type: Superiority; p = 0.961, ANOVA; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1.2 to 1.1]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for BMI-Month 6; Test type: Superiority; p = 0.581, ANOVA; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.8 to 1.5]

14. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Waist Circumference at Month 6
Description: Values for Waist Circumference are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 6 (End of Study)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 123 | 122
cm | 0 (6.4) | 0.4 (5.9)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Waist Circumference-Month 6; Test type: Superiority; p = 0.871, ANOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.7 to 3.1]

15. Secondary Outcome: Change From Baseline of Nutritional Status Determined by Protein and Calories at Month 3 and 6
Description: Values for Protein and Calories are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 91 | 87
grams
  Protein: Month 3 | -5.6 (14.1) | -4.9 (45.3)
  Protein: Month 6 | -0.1 (24.8) | 4.5 (32.9)
  Calories: Month 3 | -76.8 (316.9) | -199.1 (525.1)
  Calories: Month 6 | 30.9 (589.5) | 108 (654)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Protein-Month 3; Test type: Superiority; p = 0.608, ANOVA; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-14.7 to 25]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Protein-Month 6; Test type: Superiority; p = 0.731, ANOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-11.5 to 8.1]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Calories-Month 3; Test type: Superiority; p = 0.377, ANOVA; Mean Difference (Final Values) = 185.3, 95% CI 2-sided [-227.5 to 598.1]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Calories-Month 6; Test type: Superiority; p = 0.854, ANOVA; Mean Difference (Final Values) = -18.3, 95% CI 2-sided [-214.4 to 177.8]

16. Secondary Outcome: Change From Baseline in QOL Based pm the EQ 5D Questionnaire Index at Month 3 and 6
Description: European Quality of Life, 5 Dimensions (EQ-5D) generates a single index score based on a descriptive system that defines health in terms of 5 dimensions, consisting of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The possible range for each dimension is 1 to 3, where 1=no problems, 2=moderate problems, 3=extreme problems. Higher score implies more problems (worsening). According to this classification, 243 potential health states are defined Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
Percent Change
  Month 3 | -0.01 (0.18) | -0.04 (0.19)
  Month 6 | -0.04 (0.19) | -0.03 (0.17)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for EQ 5D Questionnaire Index-Month 3; Test type: Superiority; p = 0.412, ANOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for EQ 5D Questionnaire Index-Month 6; Test type: Superiority; p = 0.485, ANOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.03]

17. Secondary Outcome: Change From Baseline in QOL Based on the EQ 5D Quest Health Status at Month 3 and 6
Description: Visual analogue scale to generate a self-perceived rating of health status. Visual analogue scale is the second part of the questionnaire, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine". Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
Score on a Scale
  Month 3 | -2.33 (23.37) | -2.58 (27.14)
  Month 6 | -1.60 (24.02) | 0.92 (30.22)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for EQ 5D Quest Health Status-Month 3; Test type: Superiority; p = 0.525, ANOVA; Mean Difference (Final Values) = 2.18, 95% CI 2-sided [-4.56 to 8.93]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for EQ 5D Quest Health Status-Month 6; Test type: Superiority; p = 0.995, ANOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-6.79 to 6.83]

18. Secondary Outcome: Change From Baseline in QOL Based on the Diabetes Symptom Checklist (DSC) at Month 3 and 6
Description: The Diabetes Symptoms Checklist was designed to assess the presence and perceived burden of diabetes-related symptoms. Respondents were to consider troublesomeness of 34 symptoms on a 5-point scale ranging from 5="extremely" to 1="not at all." For symptoms/side-effects not experienced, the item was scored as 0. Symptoms were grouped into the following subscales: psychological fatigue, psychological cognitive, neurology pain, neurology sensory, cardiology, ophthalmology, hypoglycemia, hyperglycemia. Subscale scores were calculated as the sum of the given subscale divided by the total number of items in the scale. Total score was computed from the sum of the 8 subscales and ranged from 0 to 40. Higher scores indicate greater symptom burden. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 3, Month 6 (End of Study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 127 | 124
Scores on a scale
  Psychology, fatigue: Month 3 | 2.34 (20.73) | 2.39 (20.33)
  Psychology, fatigue: Month 6 | 2.48 (22.95) | -0.49 (24.64)
  Psychology, cognitive: Month 3 | 0.16 (18.54) | 2.66 (18.38)
  Psychology, cognitive: Month 6 | 2.23 (18.87) | 1.70 (17.23)
  Neurology, pain: Month 3 | -3.46 (17.87) | 0.32 (19.18)
  Neurology, pain: Month 6 | -1.57 (21.09) | -1.75 (22.34)
  Neurology, sensory: Month 3 | -2.25 (16.96) | 0.55 (16.09)
  Neurology, sensory: Month 6 | -0.19 (17.15) | -3.59 (15.76)
  Cardiology: Month 3 | 1.18 (17.32) | 0.87 (15.84)
  Cardiology: Month 6 | 3.60 (17.74) | 0.29 (18.11)
  Ophthalmology: Month 3 | 1.53 (21.98) | 2.24 (19.71)
  Ophthalmology: Month 6 | -0.26 (24.53) | 0.23 (19.43)
  Hypoglycemia: Month 3 | 0.49 (20.72) | 0.12 (21.02)
  Hypoglycemia: Month 6 | 0.50 (22.25) | -1.62 (21.72)
  Hyperglycemia: Month 3 | -2.07 (17.38) | -1.79 (18.83)
  Hyperglycemia: Month 6 | -0.79 (19.50) | -2.82 (18.25)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Psychology Fatigue-Month 3; Test type: Superiority; p = 0.526, ANOVA; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-7.64 to 3.91]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Psychology Fatigue-Month 6; Test type: Superiority; p = 0.779, ANOVA; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-5.01 to 6.68]
Statistical Analysis 3: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Psychology Cognitive-Month 3; Test type: Superiority; p = 0.246, ANOVA; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-7.95 to 2.04]
Statistical Analysis 4: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Psychology Cognitive-Month 6; Test type: Superiority; p = 0.780, ANOVA; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-5.78 to 4.34]
Statistical Analysis 5: Comparison: Non-Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Neurology Pain-Month 3; Test type: Superiority; p = 0.885, ANOVA; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-5.22 to 6.04]
Statistical Analysis 6: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Neurology Pain-Month 6; Test type: Superiority; p = 0.128, ANOVA; Mean Difference (Final Values) = 4.41, 95% CI 2-sided [-1.28 to 10.10]
Statistical Analysis 7: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Neurology Sensory-Month 3; Test type: Superiority; p = 0.701, ANOVA; Mean Difference (Final Values) = 1.07, 95% CI 2-sided [-4.40 to 6.54]
Statistical Analysis 8: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Neurology Sensory-Month 6; Test type: Superiority; p = 0.010, ANOVA; Mean Difference (Final Values) = 7.21, 95% CI 2-sided [1.70 to 12.73]
Statistical Analysis 9: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Cardiology-Month 3; Test type: Superiority; p = 0.934, ANOVA; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-4.63 to 5.03]
Statistical Analysis 10: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Cardiology-Month 6; Test type: Superiority; p = 0.209, ANOVA; Mean Difference (Final Values) = 3.13, 95% CI 2-sided [-1.75 to 8.01]
Statistical Analysis 11: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Ophthalmology-Month 3; Test type: Superiority; p = 0.585, ANOVA; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-4.90 to 8.68]
Statistical Analysis 12: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Ophthalmology-Month 6; Test type: Superiority; p = 0.641, ANOVA; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-5.22 to 8.47]
Statistical Analysis 13: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Hypoglycemia-Month 3; Test type: Superiority; p = 0.586, ANOVA; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-6.89 to 3.90]
Statistical Analysis 14: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Hypoglycemia-Month 6; Test type: Superiority; p = 0.906, ANOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-5.79 to 5.14]
Statistical Analysis 15: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Hyperglycemia-Month 3; Test type: Superiority; p = 0.970, ANOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-4.93 to 4.75]
Statistical Analysis 16: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Hyperglycemia-Month 6; Test type: Superiority; p = 0.340, ANOVA; Mean Difference (Final Values) = 2.38, 95% CI 2-sided [-2.52 to 7.28]

19. Secondary Outcome: Change From Baseline of MRI Body Composition at Month 6
Description: Values for Abdominal Subcutaneous Fat Volume and Abdominal Visceral Fat Volume are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 6 (End of Study)
Population: ITT of MRI sub-study (n=88 consented to participate), however, only a subset of MRI sub-study that had evaluable data were used in this analysis. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 39 | 43
mL
  Abdominal Visceral Fat Volume: Month 6: number analyzed (Participants) | 38 | 43
  Abdominal Visceral Fat Volume: Month 6 | -49 (81.7) | -64.8 (73.2)
  Abdominal Subcutaneous Fat Volume: Month 6 | -12 (58.9) | -3.3 (70.2)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Abdominal Subcutaneous Fat Volume-Month 6; Test type: Superiority; p = 0.495, ANOVA; Mean Difference (Final Values) = 24.6, 95% CI 2-sided [-46.9 to 96]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for Abdominal Visceral Fat Volume-Month 6; Test type: Superiority; p = 0.081, ANOVA; Mean Difference (Final Values) = 55.4, 95% CI 2-sided [-7 to 117.8]

20. Secondary Outcome: Change From Baseline of Left Ventricular (LV) End Diastolic and Systolic Volume as Determined by MRI at Month 6
Description: Values for Left Ventricular (LV) End Diastolic and Systolic Volume are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 6 (End of Study)
Population: ITT of MRI sub-study (n=88 consented to participate),however, only a subset of MRI sub-study that had evaluable data were used.. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 39 | 43
mL
  LV End Diastolic Volume | 2.1 (35.5) | 0.7 (28.4)
  LV End Systolic Volume | 3.3 (28.1) | -0.2 (28.4)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LV End Diastolic Volume-Month 6; Test type: Superiority; p = 0.626, ANOVA; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [-19.3 to 31.9]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LV End Systolic Volume-Month 6; Test type: Superiority; p = 0.486, ANOVA; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-14.5 to 30.1]

21. Secondary Outcome: Change From Baseline of Left Ventricular (LV) Mass Without and With Pap Muscles as Determined by MRI at Month 6
Description: Values for Left Ventricular (LV) Mass Without and With Pap Muscles are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 6 (End of Study)
Population: ITT of MRI sub-study (n=88 consented to participate), however, only a subset of MRI sub-study that had evaluable data were used.. The data in this outcome measure is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 39 | 43
grams
  LV Mass Without Pap Muscles | 0.6 (38.4) | 3.3 (26.5)
  LV Mass With Pap Muscles | 1.1 (39.2) | 3.5 (26.6)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LV Mass with Pap Muscles-Month 6; Test type: Superiority; p = 0.832, ANOVA; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-18.9 to 23.4]
Statistical Analysis 2: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LV Mass without Pap Muscles-Month 6; Test type: Superiority; p = 0.820, ANOVA; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-18.3 to 23.1]

22. Secondary Outcome: Change From Baseline of Left Ventricular (LV) Ejection Fraction as Determined by MRI at Month 6
Description: Values for Left Ventricular (LV) Ejection Fraction are included. Statistical analysis includes estimates of Least Squares (LS) comparing differences between treatment groups by visit and p-value using analysis of covariance (ANOVA) testing that the differences=0.
Time Frame: Baseline, Month 6 (End of Study)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Number analyzed (Participants) | 39 | 42
Percent | -0.3 (8.2) | 0.9 (10.4)
Statistical Analysis 1: Comparison: Non-Glucose Sparing Prescriptions vs Glucose Sparing Prescriptions; Estimate of Least Square Means Comparing Treatment Groups for LV Ejection Fraction-Month 6; Test type: Superiority; p = 0.955, ANOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-6.9 to 6.5]

ADVERSE EVENTS:
Description: The data represented in this module is a pooled analysis of the following 3 studies: NCT00567489 (protocol ID 31998), NCT00567398 (protocol ID 34202), NCT01219959 (protocol ID51067). Given that the glucose content of the PD solutions is similar, the pooling of the results were considered a valid method to answer the underlying research questions.
Arm/Group | Non-Glucose Sparing Prescriptions | Glucose Sparing Prescriptions
Serious Adverse Events (participants affected / at risk) | 41/127 | 58/124
Other Adverse Events (participants affected / at risk) | 101/127 | 98/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Glucose Sparing Prescriptions (N=127) | Glucose Sparing Prescriptions (N=124)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 2 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 2
Cardiorespiratory Arrest (Cardiac disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Heart Failure (Cardiac disorders) | 0 | 1
Ischemic Heart Disease (Cardiac disorders) | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 2 | 3
Peritonitis Associated To Peritoneal Dialysis (Gastrointestinal disorders) | 0 | 1
Peritonitis By Capd (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Catheter Related Complication (General disorders) | 2 | 1
Catheter Site Haemorrhage (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Non Specific Thoracic Pain (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Sudden Death (General disorders) | 1 | 0
Thoracic Pain (General disorders) | 1 | 0
Hypersensitivity Icodextrin (Immune system disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Abscess In Abdominal Wall (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Bacterial Peritonitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 3
Cellulitis Of Face (Infections and infestations) | 1 | 0
Cellulitis With Soft Tissue Necrosis Of The Right Hand (Infections and infestations) | 1 | 0
Entero Invasive Diarrhea (Infections and infestations) | 0 | 1
Eschar In The Left Thigh Region (Infections and infestations) | 0 | 1
Facial Abscess (Infections and infestations) | 1 | 0
Fungal Peritonitis (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Nosocomial Pneumonia (Infections and infestations) | 0 | 1
Peritonitis Bacterial (Infections and infestations) | 5 | 8
Pneumonia (Infections and infestations) | 2 | 2
Post Traumatic Cellulitis (Infections and infestations) | 0 | 1
Right Basal Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 1
Thigh Abscess (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Blood Glucose Abnormal (Investigations) | 1 | 0
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 1
Fluid Overload (Metabolism and nutrition disorders) | 3 | 5
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Severe Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 2
Neurotoxicity (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Seizures (Nervous system disorders) | 0 | 1
Sensory Impairment (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Thalamic Infarction (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Left Malleolus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Local Infection Of The Skin (Diabetic Sore) (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Blood Pressure Inadequately Controlled (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 3
Hypertensive Urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Glucose Sparing Prescriptions (N=127) | Glucose Sparing Prescriptions (N=124)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Anemia (Blood and lymphatic system disorders) | 2 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 2 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 2
Cardiorespiratory Arrest (Cardiac disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Heart Failure (Cardiac disorders) | 0 | 1
Ischemic Heart Disease (Cardiac disorders) | 1 | 0
Left Atrial Enlargement (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 2 | 1
Hyperparathyroidism Secondary (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diabetic Retinopathy (Eye disorders) | 0 | 1
Dry Eye (Eye disorders) | 2 | 0
Eye Haemorrhage (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 1 | 1
Eye Pruritus (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Myodesopsia (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Acute Diarrhea (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Bloody Peritoneal Effluent (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 8
Diabetic Gastropathy (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Epigastric Pain (Gastrointestinal disorders) | 2 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Hyperemesis (Gastrointestinal disorders) | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 6 | 4
Nauseas (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pain In Teeth (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 10 | 10
Peritonitis Associated To Peritoneal Dialysis (Gastrointestinal disorders) | 0 | 1
Peritonitis By Cap (Gastrointestinal disorders) | 1 | 0
Peritonitis By Capd (Gastrointestinal disorders) | 1 | 2
Reflux Oesophagitis (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 9
Application Site Oedema (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 4
Catheter Related Complication (General disorders) | 4 | 4
Catheter Site Discharge (General disorders) | 1 | 1
Catheter Site Haemorrhage (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Granuloma (General disorders) | 1 | 0
Granuloma In Exit-Site (General disorders) | 0 | 1
Granuloma Of The Exit Site (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Injection Site Papule (General disorders) | 1 | 0
Mild Erythema Of Catheter Exit Site (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Non Specific Thoracic Pain (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema (General disorders) | 8 | 0
Oedema Peripheral (General disorders) | 10 | 2
Peritoneal Catheter Dysfunction (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sickness (General disorders) | 1 | 1
Sudden Death (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Thoracic Pain (General disorders) | 1 | 0
Xerosis (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Hypersensitivity Icodextrin (Immune system disorders) | 0 | 1
Skin Allergic Reaction (Immune system disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Abscess In Abdominal Wall (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Bacterial Peritonitis (Infections and infestations) | 2 | 1
Candidiasis (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 5 | 5
Cellulitis (Infections and infestations) | 1 | 3
Cellulitis Of Face (Infections and infestations) | 1 | 0
Cellulitis With Soft Tissue Necrosis Of The Right Hand (Infections and infestations) | 1 | 0
Diarrhoea Infectious (Infections and infestations) | 0 | 1
Entero Invasive Diarrhea (Infections and infestations) | 0 | 1
Eschar In The Left Thigh Region (Infections and infestations) | 0 | 1
Exit Site Infection (Infections and infestations) | 1 | 1
Exit Site Infection Of Catheter (Infections and infestations) | 0 | 1
Facial Abscess (Infections and infestations) | 1 | 0
Flu (Infections and infestations) | 2 | 2
Folliculitis (Infections and infestations) | 0 | 1
Fungal Peritonitis (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Herpes Virus Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Nosocomial Pneumonia (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Peritonitis Bacterial (Infections and infestations) | 7 | 8
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2
Post Traumatic Cellulitis (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Right Basal Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 1
Severe Acute Respiratory Syndrome (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Skin Infection Staphylococcus (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 1 | 0
Thigh Abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4
Urinary Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 6 | 2
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Bitten By A Dog On The Left Leg (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Dialysis Device Complication (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Excoriation On Knees (Injury, poisoning and procedural complications) | 1 | 0
Fracture Right Leg (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 2 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 1
Trauma Of Soft Tissue (Injury, poisoning and procedural complications) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Calcium Decreased (Investigations) | 1 | 0
Blood Glucose Abnormal (Investigations) | 1 | 0
Blood Magnesium Decreased (Investigations) | 1 | 0
Blood Parathyroid Hormone Increased (Investigations) | 2 | 0
Blood Phosphorus Decreased (Investigations) | 0 | 1
Blood Urea Increased (Investigations) | 1 | 0
Decreased Peripheral Pulses (Investigations) | 0 | 1
Electrocardiogram T Wave Inversion (Investigations) | 2 | 0
Fibrin Abnormal (Investigations) | 0 | 1
Haemoglobin Increased (Investigations) | 1 | 0
Heart Murmur (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1
St Segment Depression (Investigations) | 1 | 0
T Peaked (Investigations) | 0 | 1
Urine Output Decreased (Investigations) | 1 | 0
Weight Increased (Investigations) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0
Diabetic Foot (Metabolism and nutrition disorders) | 3 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Dyslipidemia (Metabolism and nutrition disorders) | 0 | 1
Fluid Imbalance (Metabolism and nutrition disorders) | 1 | 1
Fluid Overload (Metabolism and nutrition disorders) | 6 | 8
Fluid Retention (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 3 | 1
Hypervolemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyporexia (Metabolism and nutrition disorders) | 1 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 3 | 5
Mild Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Moderate Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Severe Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower Limbs Cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Bilateral Legs (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Right Knee Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Carcinoid Tumour Of The Duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burning Sensation (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Diabetic Encephalopathy (Nervous system disorders) | 1 | 0
Diabetic Neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 3
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 3
Hypoesthesia Hands And Feet (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Seizures (Nervous system disorders) | 0 | 1
Sensory Impairment (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Thalamic Infarction (Nervous system disorders) | 0 | 1
Third Cranial Nerve Neuropathy (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 4
Sadness (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 3 | 0
Exfoliative Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypopigmented Skin Lesions (Skin and subcutaneous tissue disorders) | 0 | 1
Left Malleolus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Local Infection Of The Skin (Diabetic Sore) (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 0 | 1
Dialysis (Surgical and medical procedures) | 1 | 0
Accelerated Hypertension (Vascular disorders) | 1 | 0
Arterial Hypertension (Vascular disorders) | 0 | 1
Arterial Stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis Obliterans (Vascular disorders) | 1 | 0
Blood Pressure Inadequately Controlled (Vascular disorders) | 1 | 0
Diabetic Vascular Disorder (Vascular disorders) | 1 | 0
Digital Ischemia In The 1st And 2nd Of The Feet (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 6
Hypertensive Crisis (Vascular disorders) | 1 | 3
Hypertensive Urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 2
Ischaemia (Vascular disorders) | 1 | 0
Jugular Vein Distension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This is a pooled analysis of NCT00567489, NCT00567398, and NCT01219959. Given that the glucose content of the PD solutions were similar, the pooling of the results were considered a valid method to answer the underlying research questions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes